CLINICAL TRIAL: NCT01322243
Title: Effect of Metabolic State on Anxiety in Human Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to mechanical issue with device
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EKE-0724
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Volunteers
Keywords: Anxiety; Metabolic state; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Intervention: Fasted State (Other): Participants will be randomized to a dietary intervention of a fasted or fed group upon admission.
  Interventions: Other: Dietary manipulation
- Dietary Intervention: Fed State (Other): Participants will be randomized to a dietary intervention of a fasted or fed group upon admission
  Interventions: Other: Dietary manipulation

INTERVENTIONS:
Other: Dietary manipulation — Participants are maintained in a fasted (only noncaloric beverages) or fed (isocaloric weight-maintenance diet) state for two days.

SUMMARY:
In this study, we would like to explore the hypothesis that changes in metabolic state, induced by altering hormone levels and patterns of neural activity, affect the experience of anxiety in humans. We will also investigate if there is a link between high anxiety and higher caloric intake. Our aim is to characterize whether changes in current metabolic state systematically influence anxiety induced by a well established behavioral task known as the threat of shock. The neural regions activated by this behavioral task in healthy subjects have been well characterized. We have a priori regions of interest that include the insula, anterior cingulate cortex, hypothalamus, amygdala, and prefrontal cortex. As our primary outcome, we will assess neural activation with whole-brain functional magnetic resonance imaging to determine whether brain regions are differentially engaged when subjects experience anxiety across different metabolic states. We will correlate these changes with psychophysiological measures of anxiety and metabolic state.

DETAILED DESCRIPTION:
There is evidence that our subjective experience of the world is strongly influenced by our metabolic state, the status of our body's energy reserves and level of hunger. Hormones that regulate appetite, food ingestion and body weight apparently also exert their action on neuroanatomical circuits involved in the generation of psychological states. Previous research indicates that an individual's metabolic state may influence their susceptibility to and experience of anxiety. Conversely, stress can also modulate appetite and body weight regulation. There are many clinical implications of the bidirectional relationship between stress/anxiety and metabolic state/energy regulation but two of the most important ones are obesity and eating disorders. In terms of obesity, the high recidivism after successful weight loss underscores the limited use of caloric restriction to treat obesity. It is unknown whether dieting (fasting) increases anxiety, which eventually may undermine an individual's motivation to restrict food intake. Research shows that anxiety can increase appetite and exacerbate the physical and psychological manifestations associated with hunger. However, there is a paucity of experimental data establishing whether the metabolic changes associated with fasting influence the experience of stress and possibly, an individual's ability to continue dieting for an extended period of time. In the setting of both obesity and anorexia nervosa, the levels of metabolic hormones are different to those found in people of normal body weight. It is therefore likely that the activation of brain regions associated with energy and body weight regulation is abnormal. Many of these brain regions are also involved in the control of anxiety responses. The fact that there is a high comorbidity between anorexia nervosa and anxiety disorders indicates the potential contribution of metabolic states to the perception of stress.

To better understand the relationship between metabolic state and anxiety, we will examine whether changes in metabolic state influence anxiety in human subjects. We will use whole-brain functional magnetic resonance imaging (fMRI) to identify the neural mechanisms that underlie metabolic state-dependent changes in the response to anxiety-inducing stress. In a randomized crossover design, participants will be tested in a well-established behavioral task that elicits anticipatory anxiety in two separate sessions that differ with respect to their metabolic states. We aim to perform a fine-grain analysis of changes in neural and physiological responses to this anxiety-inducing task as a function of metabolic state. Using fMRI as well as non-invasive psychophysiological measures, we will characterize whether there are systematic differences in the neural and psychophysiological experience of anxiety across different metabolic states in obese as compared to lean individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 - 40 years.
* Body Mass Index (BMI) from 19.0 to 25.0 for the lean population or Body Mass Index (BMI) equal to or greater than 30 for the obese population and under 300lbs (136.07kg.)
* Fluent in English
* Females must report a normal menstrual cycle length defined as from 24-35 days, with a period lasting from 2-7 days
* Stable weight (+/- 5 %) for at least three months prior to each admission and under 300 lbs (136.07kg.)

Exclusion Criteria:

* Weight of > 300 lbs (136.07kg.)
* Patients may not have had > 550 mL of blood drawn within 8 weeks of study entry.
* Less than 8 weeks after receiving an investigational new drug (IND). Patients must have a minimum of an 8 week washout period.
* Left-handedness.
* Any employee of Rockefeller University who knows the details of this study
* Reported history of claustrophobia.
* Reported history of metal implants, pacemaker, IUD, braces, or tattoos less then 6 months old.
* Reported history of smoking, chewing tobacco or use of nicotine patches within the previous 3 months.
* Reported history of alcohol abuse/dependence.
* Reported use of prescription medication for pain, anxiety or sleep more than once a week.
* Reported daily ingestion of herbal (including melatonin) or dietary supplements within one month prior to the screening.
* Reported use of medications or herbal supplements that affect appetite or body weight within the previous three months.
* Reported history of using the following medications: glucocorticoids, anti-seizure medications, thyroid hormones in the past six months.
* Reported Psychiatric disorder requiring medication or treatment.
* Reported history of cardiac disease.
* Reported history of illnesses that affect metabolic hormone levels: renal or hepatic failure, type 1 or type 2 diabetes, lymphoma, hypogonadism, malabsorption/malnourishment, hypo- or hyper-thyroidism, hypercortisolism or any endocrinopathies.
* Reported history of physical exercise >2 hours per day.
* Reported history by female subjects of amenorrhea (no periods for longer than 3 months (even with negative uhCG) and oligomenorrhea (length greater than 35 days.)
* Pregnant (verified by urine hCG) or breast-feeding within the past 3 months.
* Eating disorder as suggested by at least 2 'yes' answers on the SCOFF Eating Disorder Questionnaire.
* Alcohol dependence as suggested by at least 2 'yes' answers on the CAGE Questionnaire.
* Current use of any illicit drug (including "recreational use") as verified by urine toxicology test.
* Anemia defined as Hgb < 12g/dL for male subjects < 11g/d/L for female subjects.
* TSH level that is outside the reference range of 0.3 - 0.5 mU/L or free T4 level that is outside the reference range of 4.5 - 11.2 mcg/dL (performed only if an abnormal thyroid gland identified on physical examination.)
* History, physical, social or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI, make the candidate ineligible for the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) blood oxygenation level dependent (BOLD) signals as indications of neural activity during exposure to an anxiety-inducing stress. | 4 years

SECONDARY OUTCOMES:
Physiological and behavioral parameters of emotional and metabolic state. | 4 years
  Physiologic and behavioral assessment:
  Metabolic state:
  * Hormone levels will be obtained every morning during the two days of fasting or normal food consumption
  * Subjective measures of metabolic state will be accomplished through the use of the hunger questionnaire and the hunger visual analog scale.
  * Body composition will be obtained on the first and last days of admission.
  * Food consumption measured in calories immediately after the fMRI experiment.
  Anxiety state:
  * Salivary cortisol tests will be performed
  * Physiological measures of anxiety, in addition to plasma ACTH, salivary cortisol testing, plasma epinephrine and norepinephrine
  * Emotional status will be evaluated through the use of the questionnaires
Response inhibition (impulse control) is also a secondary outcome for this study | 4 years
  Impulse control will be assessed with the validated cognitive task

CONTACTS AND LOCATIONS:
Overall Officials: Ana Emiliano, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States